CLINICAL TRIAL: NCT01226394
Title: Multicentric Phase III Trial Comparing Simple Follow-up to Exploratory Laparotomy Plus "in Principle" HIPEC (Hyperthermic Intraperitoneal Chemotherapy) in Colorectal Patients Initially Treated With Surgery and Adjuvant Chemotherapy Who Have a High Risk of Developing Colorectal Peritoneal Carcinomatosis
Brief Title: Trial Comparing Simple Follow-up to Exploratory Laparotomy Plus "in Principle" (Hyperthermic Intraperitoneal Chemotherapy) HIPEC in Colorectal Patients
Acronym: ProphyloCHIP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSET 1539-ProphyloCHIP; 2009-015598-11 (EudraCT Number)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer With a Resected Minimal Synchronous PC; Ovarian Metastases; Tumour Rupture in the Abdominal Cavity
Keywords: peritoneal carcinomatosis; HIPEC; controlled clinical trial
MeSH Terms: conditions — Krukenberg Tumor; Peritoneal Neoplasms | interventions — Laparotomy; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surveillance (No Intervention)
- laparotomy plus HIPEC. (Experimental)
  Interventions: Procedure: laparotomy plus HIPEC

INTERVENTIONS:
Procedure: laparotomy plus HIPEC — Laparotomy + HIPEC
  Arms: laparotomy plus HIPEC.

SUMMARY:
Multicentric randomised trial. Patients with a high risk of developing colorectal Peritoneal Carcinomatosis (PC) after resection of their primary will be informed, will sign the consent and will be pre-registered. All patients will receive the current standard adjuvant treatment : 6 months of systemic chemotherapy (currently the Folfox-4 regimen which could be modified if the standard is modified). Then a work-up is done to exclude recurrence. The likelihood of a recurrence is low but if this occurs, the patient will not be randomised and will be treated with the best known treatment. If the work-up is negative, patients will be randomised to surveillance alone (control group) or exploratory laparotomy + HIPEC (experimental group).

ELIGIBILITY:
Inclusion Criteria:

A) Patients presenting with the following history:

1. Histologically-proven colorectal adenocarcinoma
2. Presenting at the time of resection of the primary with one of the following 4 criteria (criteria indicating a high risk of developing PC) :

   * Minimal PC, resected at the same time as the primary
   * Ovarian metastases
   * Rupture of the primary tumour inside the peritoneal cavity,
   * Iatrogenic rupture of the primary tumour during surgery

B) Who have received standard systemic adjuvant chemotherapy (6 months of systemic chemotherapy) :

* Chemotherapy with the Folfox 4 regimen (the current standard treatment ; it can be modified in the future in the two groups, if the standard is modified…).
* Given on an intent-to-treat basis (it can be stopped prematurely for miscellaneous reasons…);

C) Patients who do not present any sign of tumour recurrence at the end of these 6 months of chemotherapy.

D) Patients with the following general characteristics:

1. Age between 18 and 70 years,
2. Performance Status WHO < 2, life expectancy > 12 weeks,
3. Haematological parameters : Polynuclear neutrophils ³ 1.5x109/L, platelets ³ 100x109/L,
4. Liver function : Total Bilirubin £ 1.5 x ULN, AST (SGOT) et ALT (SGPT) £ 3 x ULN, alkaline phosphatases £ 3 x ULN,
5. Renal function : Plasma creatinine £ 1,25 x ULN,
6. Operable patients,
7. Grade £ 2 peripheral neuropathy (CTC AE v3.0 annex 7)
8. Patients entitled to French National Health Insurance coverage.

E)Patients will be informed and a signed consent form will be obtained before initiating any procedure specific to the trial.

Exclusion Criteria:

1. Cancers of non colorectal origin, particularly, appendiceal cancers are excluded
2. Patients presenting with a detectable recurrent tumour
3. Grade ≥ 3 Peripheral neuropathy
4. History of cancer (excepted cutaneous basocellullar cancer or in situ carcinoma of the uterine cervix) with a recurrence during the 5 previous years
5. Patients already included in another trial concerning first-line treatment 6) Pregnant women or likely to be pregnant

7) Persons under guardianship 8) Follow-up impossible for geographic, social or psychological reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-04; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To increase the 3-year disease-free survival | 3 years
  3-year disease-free survival

SECONDARY OUTCOMES:
3 year overall survival | 3 years
Peritoneal disease-free survival | 3 years
5 year overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Diane GOERE, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Goere D, Glehen O, Quenet F, Guilloit JM, Bereder JM, Lorimier G, Thibaudeau E, Ghouti L, Pinto A, Tuech JJ, Kianmanesh R, Carretier M, Marchal F, Arvieux C, Brigand C, Meeus P, Rat P, Durand-Fontanier S, Mariani P, Lakkis Z, Loi V, Pirro N, Sabbagh C, Texier M, Elias D; BIG-RENAPE group. Second-look surgery plus hyperthermic intraperitoneal chemotherapy versus surveillance in patients at high risk of developing colorectal peritoneal metastases (PROPHYLOCHIP-PRODIGE 15): a randomised, phase 3 study. Lancet Oncol. 2020 Sep;21(9):1147-1154. doi: 10.1016/S1470-2045(20)30322-3. Epub 2020 Jul 24. PMID 32717180
- See also: Related Info — http://igr.fr